CLINICAL TRIAL: NCT05942885
Title: Hypnosis: a Path to Appeasement
Acronym: HYCVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL23_0336
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Cancer
Keywords: hypnosis; Diffuse large cell B-cell lymphoma; follicular lymphoma; anxiety
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anxiety scores (Experimental)
  Interventions: Other: anxiety questionnaire

INTERVENTIONS:
Other: anxiety questionnaire — Patient undergoing hypnosis session will have their anxiety measured just before the third session of hypnosis and after during a telephonic consultation. The result will be compared to the anxiety level before the first hypnosis session

SUMMARY:
Hypnosis is a technique allowing the patient to focus his mental attention on a thought or a sensation, with the aim of reducing or modulating the intensity of a negative feeling or an ordeal encountered during the course of treatment. This tool can be used when patients are faced with chronic disorders (pain, anxiety, ...) or iatrogenic effects (nausea, asthenia, ...).

The patient is referred to hypnosis care by the doctor, psychologist or paramedics who follow him, when they detect a need.

Several scientific studies have shown the effectiveness of hypnosis in improving the quality of life of patients with breast cancer and in reducing pain during invasive procedures. On the other hand, in hematology, no research has measured the evolution of anxiety, over time, in patients receiving hypnotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, fluent in French.
* Patients starting hypnotherapy for anxiety disorders.
* Anxiety score on the HADS scale (Hospital Anxiety and Depression Scale) greater than or equal to 8/21
* Patients with diffuse large cell B-cell lymphoma or follicular lymphoma, whatever the stage of the disease.
* Diagnosis announcement less than 2 months old

Exclusion Criteria:

* Persons deprived of their liberty by a judicial or administrative decision
* Adults subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of anxiety | Week 6 after 2 hypnosis sessions
  Difference in anxiety measured before starting hypnotherapy care and after 2 hypnosis sessions. It will be measured by the Hospital Anxiety and Depression Scale. This scale gives a score according to the level of anxiety ranging from 0 to 21. The higher the score, the more the patient is anxious.

SECONDARY OUTCOMES:
Evolution of anxiety before hypnotherapy and after 3 months of follow-up in hypnotherapy | Month 3 after 3 hypnosis sessions
  Difference in anxiety measured before starting hypnotherapy care and after 3 hypnosis sessions. It will be measured by the Hospital Anxiety and Depression Scale. This scale gives a score according to the level of anxiety ranging from 0 to 21. The higher the score, the more the patient is anxious.
Evolution of anxiety between D0 and M3 according to the type of lymphoma | Month 3 after 3 hypnosis sessions
  Difference in anxiety measured before starting hypnotherapy care and after 3 hypnosis sessions for two subgroups : follicular lymphoma and diffuse large b-cell lymphoma. It will be measured by the Hospital Anxiety and Depression Scale. This scale gives a score according to the level of anxiety ranging from 0 to 21. The higher the score, the more the patient is anxious.
Evolution of anxiety between D0 and W6 according to the type of lymphoma | Week 6 after 2 hypnosis sessions
  Difference in anxiety measured before starting hypnotherapy care and after 2 hypnosis sessions for two subgroups : follicular lymphoma and diffuse large b-cell lymphoma. It will be measured by the Hospital Anxiety and Depression Scale. This scale gives a score according to the level of anxiety ranging from 0 to 21. The higher the score, the more the patient is anxious.
Evolution of anxiety between D0 and W6 according to the gender of the patient | Week 6 after 2 hypnosis sessions
  Difference in anxiety measured before starting hypnotherapy care and after 2 hypnosis sessions for two subgroups : man and woman. It will be measured by the Hospital Anxiety and Depression Scale. This scale gives a score according to the level of anxiety ranging from 0 to 21. The higher the score, the more the patient is anxious.
Evolution of anxiety between D0 and M3 according to the gender of the patient | Month 3 after 3 hypnosis sessions
  Difference in anxiety measured before starting hypnotherapy care and after 3 hypnosis sessions for two subgroups : man and woman. It will be measured by the Hospital Anxiety and Depression Scale. This scale gives a score according to the level of anxiety ranging from 0 to 21. The higher the score, the more the patient is anxious.
Evolution of anxiety between D0 and W6 according to age category | Week 6 after 2 hypnosis sessions
  Difference in anxiety measured before starting hypnotherapy care and after 2 hypnosis sessions for two subgroups : under 60 years old ans over 60 years old. It will be measured by the Hospital Anxiety and Depression Scale. This scale gives a score according to the level of anxiety ranging from 0 to 21. The higher the score, the more the patient is anxious.
Evolution of anxiety between D0 and M3 according to age category | Month 3 after 3 hypnosis sessions
  Difference in anxiety measured before starting hypnotherapy care and after 3 hypnosis sessions for two subgroups : under 60 years old ans over 60 years old. It will be measured by the Hospital Anxiety and Depression Scale. This scale gives a score according to the level of anxiety ranging from 0 to 21. The higher the score, the more the patient is anxious.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BERT, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service MB1 - Hôpital Lyon Sud - HCL, Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No